CLINICAL TRIAL: NCT06431074
Title: Radicle Calm™ 24: A Randomized, Double-Blind, Placebo-Controlled Direct-to-Consumer Study Assessing the Impact of Health and Wellness Products on Feelings of Anxiety and Related Health Outcomes
Brief Title: Radicle Calm 24: A Study of Health and Wellness Products on Feelings of Anxiety and Related Health Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radicle Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RADX-P-2402
Record Dates: First submitted 2024-05-17; First posted 2024-05-28 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Anxiety; Stress
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be stratified based on gender at birth, then randomized to one of the study arms
Who Masked: Participant, Investigator
Masking Description: The investigator is blinded to the participants' study product assignment. Participants are blinded to the study product they are assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo Control 1 (Placebo Comparator): Calm Product Form 1 - control
  Interventions: Dietary Supplement: Placebo Control Form 1
- Active Product 1.1 (Experimental): Calm Product Form 1 - active product 1
  Interventions: Dietary Supplement: Calm Active Study Product 1.1 Usage
- Placebo Control 6.1.0 (Placebo Comparator): Calm Product 6.1 - control
  Interventions: Dietary Supplement: Placebo Control 6.1
- Active Product 6.1.1 (Experimental): Calm Product 6.1 - active product 1
  Interventions: Dietary Supplement: Calm Active Study Product 6.1 Usage

INTERVENTIONS:
Dietary Supplement: Placebo Control Form 1 — Participants will use their Placebo Control Form 1 as directed for a period of 6 weeks.
  Arms: Placebo Control 1
Dietary Supplement: Calm Active Study Product 1.1 Usage — Participants will use their Radicle Calm Active Study Product 1.1 as directed for a period of 6 weeks.
  Arms: Active Product 1.1
Dietary Supplement: Placebo Control 6.1 — Participants will use their Placebo Control 6.1 as directed for a period of 6 weeks.
  Arms: Placebo Control 6.1.0
Dietary Supplement: Calm Active Study Product 6.1 Usage — Participants will use their Radicle Calm Active Study Product 6.1 as directed for a period of 6 weeks.
  Arms: Active Product 6.1.1

SUMMARY:
A randomized, double-blind, placebo-controlled study assessing the impact of health and wellness products on feelings of anxiety and related health outcomes

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study conducted with adult participants, residing in the United States.

Eligible participants will (1) endorse a desire for less feelings of anxiety (2) have the opportunity for meaningful improvement (at least 30%) in their primary health outcome, and (3) express acceptance in taking a product and not knowing its formulation until the end of the study.

Participants that report a known cardiac dysfunction, liver or kidney disease may be excluded. Participants that report a known contraindication or with well-established, significant safety concerns due to illness will be excluded. Heavy drinkers and those who report they are pregnant, trying to become pregnant, or breastfeeding will be excluded. Participants that report taking medications with a known contraindication or with well-established, significant safety concerns will be excluded.

Self-reported data are collected electronically from eligible participants over 7 weeks. Participant reports of health indicators will be collected at baseline, throughout the active period of study product use, and in a final survey. All study assessments will be electronic; there are no in-person visits or assessments for this real-world evidence study.

ELIGIBILITY:
Inclusion Criteria:

* Adults, at least 21 years of age and older at the time of electronic consent, inclusive of all ethnicities, races, genders and/or gender identities. Assigned sex at birth will determine sex-specific recruitment and surveys (male vs female) employed, when needed
* Resides in the United States
* Endorses less anxiety as a primary desire
* Has the opportunity for at least 20% improvement in their primary health outcome
* Expresses a willingness to take a study product and not know the product identity (active or placebo) until the end of the study

Exclusion Criteria:

* Reports being pregnant, trying to become pregnant, or breastfeeding
* Unable to provide a valid US shipping address and mobile phone number
* Reports current enrollment in another clinical trial
* Reports being a heavy drinker (defined as drinking 3 or more alcoholic beverages per day)
* Unable to read and understand English
* Reports a current and/or recent (up to 3 months ago) major illness and/or surgery that poses a known, significant safety risk.
* Reports a diagnosis of cardiac dysfunction, liver or kidney disease that presents a known contraindication and/or a significant safety risk with any of the study product ingredients. NYHA (New York Heart Association) Class Ill or IV congestive heart failure, atrial fibrillation, uncontrolled arrhythmias, cirrhosis, end-stage liver disease, stage 3b or 4 chronic kidney disease, or kidney failure
* Reports taking medications that have a well-established moderate or severe interaction, posing a substantial safety risk with any of the study product ingredients. Anticoagulants, antihypertensive, anxiolytics, antidepressants, chemotherapy, immunotherapy, sedative hypnotics, seizure medications, medications that warn against grapefruit consumption, corticosteroids at doses greater than 5 mg per day, diabetic medications, oral anti-infectives (antibiotics, antifungals, antivirals) to treat an acute infection, antipsychotics, MAOls (monoamine oxidase inhibitors), or thyroid products
* Reports current use of the primary ingredient(s) and/or similar product(s) to the active study product(s)
* Lack of reliable daily access to the internet

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 502 (Actual)
Dates: Start 2024-05-30 (Actual); Primary Completion 2025-08-04 (Actual); Study Completion 2025-08-11 (Actual)

PRIMARY OUTCOMES:
Change in feelings of anxiety | 6 weeks
  Mean difference in feelings of anxiety score as assessed by Patient Reported Outcome Measurement System (PROMIS) Anxiety 8A (scale 8-40; where lower scores correspond to less feelings of anxiety)

SECONDARY OUTCOMES:
Change in stress | 6 weeks
  Mean difference in stress score as assessed by Perceived Stress Scale 4 (PSS-4) (scale 0-16; where lower scores correspond to less stress)
Change in sleep | 6 weeks
  Mean difference in sleep score as assessed by Patient Reported Outcome Measurement System (PROMIS) Sleep Disturbance 4A (scale 4-20; where lower scores correspond to better sleep quality/less sleep disturbance)
Change in mood (emotional distress) | 6 weeks
  Mean difference in mood score as assessed by Patient Reported Outcome Measurement System (PROMIS) Emotional Distress-Depression 4A (scale 4-20; where lower scores correspond to lower levels of emotional distress)
Minimal clinically important difference (MCID) in feelings of anxiety | 6 weeks
  Likelihood of achieving a MCID in sleep disturbance, as measured by Patient Reported Outcome Measurement System (PROMIS) Anxiety 8A (scale 8-40; where lower scores correspond to less feelings of anxiety)
Minimal clinically important difference (MCID) in stress | 6 weeks
  Likelihood of experiencing minimal clinically important difference in stress score as assessed by Perceived Stress Scale 4 (PSS-4) (scale 0-16; where lower scores correspond to less stress)
Minimal clinically important difference (MCID) in sleep | 6 weeks
  Likelihood of experiencing minimal clinically important difference in sleep score as assessed by Patient Reported Outcome Measurement System (PROMIS) Sleep Disturbance 4A (scale 4-20; where lower scores correspond to better sleep quality/less sleep disturbance)
Minimal clinically important difference (MCID) in mood (emotional distress) | 6 weeks
  Likelihood of experiencing minimal clinically important difference in mood score as assessed by Patient Reported Outcome Measurement System (PROMIS) Emotional Distress-Depression 4A (scale 4-20; where lower scores correspond to lower levels of emotional distress)

OTHER OUTCOMES:
Change in saliva concentration of at-home (direct-to-consumer) specimen assay (1) | 6 weeks
  Mean difference in saliva concentration as assessed by saliva-based IgG (Immunoglobulin) biomarker. (Optional; among consented participants only).
Change in saliva concentration of at-home (direct-to-consumer) specimen assay (2) | 6 weeks
  Mean difference in saliva concentration as assessed by saliva-based cytokines (Interleukin 1 beta, Interleukin 8, Tumor necrosis factor-alpha, and Interleukin 6) biomarker. (Optional; among consented participants only).
Change in saliva concentration of at-home (direct-to-consumer) specimen assay (3) | 6 weeks
  Mean difference in saliva concentration as assessed by saliva-based dehydroepiandrosterone sulfate (DHEA-S) biomarker. (Optional; among consented participants only).
Change in saliva concentration of at-home (direct-to-consumer) specimen assay (4) | 6 weeks
  Mean difference in saliva concentration as assessed by saliva-based estradiol biomarker. (Optional; among consented participants only).
Change in saliva concentration of at-home (direct-to-consumer) specimen assay (5) | 6 weeks
  Mean difference in saliva concentration as assessed by saliva-based progesterone biomarker. (Optional; among consented participants only).
Change in saliva concentration of at-home (direct-to-consumer) specimen assay (6) | 6 weeks
  Mean difference in saliva concentration as assessed by saliva-based testosterone biomarker. (Optional; among consented participants only).
Change in saliva concentration of at-home (direct-to-consumer) specimen assay (7) | 6 weeks
  Mean difference in saliva concentration as assessed by saliva-based cortisol biomarker. (Optional; among consented participants only).
Change in saliva concentration of at-home (direct-to-consumer) specimen assay (8) | 6 weeks
  Mean difference in saliva concentration as assessed by saliva-based melatonin biomarker. (Optional; among consented participants only).
Change in saliva concentration of at-home (direct-to-consumer) specimen assay (9) | 6 weeks
  Mean difference in saliva concentration as assessed by saliva-based C-Reactive Protein (CRP) biomarker. (Optional; among consented participants only).
Change in blood concentration of at-home (direct-to-consumer) specimen assay (1) | 6 weeks
  Mean difference in blood concentration as assessed by blood-based cortisol biomarker (1 drop). (Optional; among consented participants only).
Change in blood concentration of at-home (direct-to-consumer) specimen assay (2) | 6 weeks
  Mean difference in blood concentration as assessed by blood-based homocysteine biomarker (1 drop). (Optional; among consented participants only).
Change in blood concentration of at-home (direct-to-consumer) specimen assay (3) | 6 weeks
  Mean difference in blood concentration as assessed by blood-based ferritin biomarker (1 drop). (Optional; among consented participants only).
Change in blood concentration of at-home (direct-to-consumer) specimen assay (4) | 6 weeks
  Mean difference in blood concentration as assessed by blood-based thyroid stimulating hormone (TSH) biomarker (1 drop). (Optional; among consented participants only).
Change in blood concentration of at-home (direct-to-consumer) specimen assay (5) | 6 weeks
  Mean difference in blood concentration as assessed by blood-based hemoglobin A1C (HbA1c) biomarker (1 drop). (Optional; among consented participants only).
Change in blood concentration of at-home (direct-to-consumer) specimen assay (6) | 6 weeks
  Mean difference in blood concentration as assessed by blood-based insulin biomarker (1 drop). (Optional; among consented participants only).
Change in blood concentration of at-home (direct-to-consumer) specimen assay (7) | 6 weeks
  Mean difference in blood concentration as assessed by blood-based vitamin D biomarker (1 drop). (Optional; among consented participants only).
Change in blood concentration of at-home (direct-to-consumer) specimen assay (8) | 6 weeks
  Mean difference in blood concentration as assessed by blood-based dehydroepiandrosterone sulfate (DHEA-S) biomarker (1 drop). (Optional; among consented male participants only).
Change in blood concentration of at-home (direct-to-consumer) specimen assay (9) | 6 weeks
  Mean difference in blood concentration as assessed by blood-based testosterone biomarker (1 drop) (Optional; among consented male participants only).
Change in blood concentration of at-home (direct-to-consumer) specimen assay (10) | 6 weeks
  Mean difference in blood concentration as assessed by blood-based estradiol biomarker (1 drop). (Optional; among consented participants only).
Change in blood concentration of at-home (direct-to-consumer) specimen assay (11) | 6 weeks
  Mean difference in blood concentration as assessed by blood-based follicle-stimulating hormone (FSH) biomarker (1 drop). (Optional; among consented female participants only).
Change in blood concentration of at-home (direct-to-consumer) specimen assay (12) | 6 weeks
  Mean difference in blood concentration as assessed by blood-based total cholesterol (high-density lipoproteins (HDL) and low-density lipoproteins (LDL)) biomarker (1 drop). (Optional; among consented participants only).
Change in blood concentration of at-home (direct-to-consumer) specimen assay (13) | 6 weeks
  Mean difference in blood concentration as assessed by blood-based triglycerides (apolipoprotein A1 (ApoA1) and apolipoprotein B (ApoB)) (1 drop). (Optional; among consented participants only).
Change in stool concentration of at-home (direct-to-consumer) specimen assay | 6 weeks
  Mean difference in stool concentration as assessed by a stool sample (microbial diversity) (Optional; among consented participants only).

CONTACTS AND LOCATIONS:
Overall Officials: Emily K. Pauli, PharmD, Principal Investigator — Radicle Science Inc.
Locations (1):
- Radicle Science, Inc, Del Mar, California, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared with researchers outside of Radicle Collaborators on this study.

REFERENCES:
- See also: Radicle Science, Inc — http://radiclescience.com